CLINICAL TRIAL: NCT06567951
Title: Maternal Supraphysiological Hypercholesterolemia: Extra Virgin Olive Oil as a Nutritional Intervention During Pregnancy to Reduce the Impact of This Maternal Condition
Brief Title: Extra Virgin Olive Oil Supplementation in Pregnancies With Increased Cholesterol Levels
Acronym: MaterLIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Universidad San Sebastián (Other)
Responsible Party: Principal Investigator, Andrea Leiva, Principal Investigator, Universidad San Sebastián
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Fondecyt 1230527
Record Dates: First submitted 2024-08-01; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy Related; Hypercholesterolemia
Keywords: Pregnancy; Cholesterol; Vascular function; Lipoprotein function; Extra virgin olive oil
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Detaile design was described in "Study Description" section. In brief: MPH and MSPH will be (or not) daily supplemented with 36 ml of EVOO from gestational week 28 to the end of pregnancy.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (without EVOO supplementation) (No Intervention): No intervention will be performed in this group of participants
- EVOO group (with EVOO supplementation) (Experimental): The intervention will be daily EVOO suplementation (36mL) form gestational week 28 until delivery
  Interventions: Dietary Supplement: Extra Virgin Olive Oil (EVOO)

INTERVENTIONS:
Dietary Supplement: Extra Virgin Olive Oil (EVOO) — This is the first time that prengnt women with maternal supraphysiological hypercholesterolemia will be suplemented with EVOO during pregnancy. The intervention will be daily EVOO suplementation (36mL) form gestational week 28 until delivery
  Arms: EVOO group (with EVOO supplementation)

SUMMARY:
The objective of this clinical trial is to know if supplementation with extra virgin olive oil (EVOO) during pregnancy, improves the maternal and neonatal lipoprotein profile, lipoprotein function, oxidative status and vascular dysfunction markers in pregnancies with maternal supraphysiological hypercholesterolemia (MSPH).

The main questions to be answered are:

1. Does 12 weeks of EVOO supplementation improve lipid and vascular outcomes in MSPH women at the end of pregnancy?
2. Does 12 weeks of EVOO supplementation improve lipid and vascular outcomes in MSPH neonates at the end of pregnancy? The investigators will compare regular diet supplemented with EVOO vs. intake of a non-supplemented regular diet to determine if EVOO reduces impaired vascular and lipid outcomes in the mother and her newborn.

Participants:

The recruited pregnant women will eat their normal diet (control group) or the same diet supplemented with 36 mL of EVOO daily (EVOO group). The protocol will be carried out from gestational week 28 to the end of pregnancy.

A nutritional specialist will evaluate every 4 weeks the EVOO consumption through surveys developed through a zoom interview.

The recruited pregnant women will have the regular obstetric control every 4 weeks.

At delivery, a maternal sample of blood as well as umbilical cord blood and the placenta will be obtained for experimental analysis.

DETAILED DESCRIPTION:
HYPOTHESIS: The nutritional supplementation with extra virgin olive oil (EVOO) enriched in polyphenols will improve the lipoprotein profile, the oxidative status and the vascular dysfunction in the mother and the offspring affected by maternal supraphysiological hypercholesterolemia (MSPH).

AIM: To determine the effects of the nutritional supplementation with EVOO during pregnancy on MSPH women, evaluating the lipoprotein profile, lipoprotein function, the oxidative status, and markers of vascular function in the mother and the offspring at birth.

STUDY DESIGN: This is a prospective, longitudinal study that aims to recruit women from week 24th (at moment where most pathological conditions of pregnancy has been diagnosed) to week 27th of gestation. These women will be supplemented with EVOO from the week 28th until term (~12 weeks). Previous studies have established that EVOO supplementation from week 28th until term reduced inflammatory markers in in pregnant women whit gestational diabetes mellitus. An equivalent group of women without EVOO supplementation will be considered as control. The participants will be from the Clínica Universidad de Los Andes (CUA). Recruitment and follow up: Pregnant women that fulfill eligibility according to the inclusion/exclusion criteria will be invited to participate in this study. They will be informed of the details of the study and will be asked to sign an informed consent for the nutritional supplementation and the biological samples donation at end of pregnancy. MPH (pregnancies with maternal physiological hypercholesterolemia or control pregnancies) or MSPH (pregnancies with maternal supraphysiological hypercholesterolemia or pathological pregnancies) will be classified at term of pregnancy according to blood TC levels, obtained by qualified personal of the Department of Obstetrics and Gynecology at CUA, under advisor of the Co- Investigator Dr. Illanes. Study groups: 1) MPH, 2) MPH + EVOO, 3) MSPH and 4) MSPH + EVOO. Inclusion criteria: pregnant women with MPH or MSPH pregnancies, with term pregnancies (≥37-weeks), singleton pregnancies, without fetal malformations, will be considered. Pregnant women with blood TC levels ≤280 mg/dl will be classified as MPH and with TC levels >280 mg/dl will be classified as MSPH. This classification is based on the criteria reported in previous published studies.

Exclusion criteria: Patients with pre-gestational and/or gestational diabetes mellitus, obesity before or during pregnancy or those with pathological conditions (e.g., pre-eclampsia, pregnancy hypertensive syndrome, and growth retardation) will be excluded from the study.

SUPPLEMENTATION: The investigators will supplement the selected women with or without EVOO since week 28th of gestation. However, the classification as MPH or MSPH occur only at birth (≥37-weeks). According to sample size calculation, the estimated sample size is 18 subjects per group. Thus 18 MSPH women supplemented with EVOO and 18 MSPH women not supplemented are required. Considering that MSPH occurs in approximately 32% of the pregnant women (data form the literature), to obtain 36 MSPH women the investigators propose to recruit 120 women in total. Thus, from these 120 women is expected that 36 will be MSPH. The other 84 women will be MPH and will be considered as control of the MSPH women. The 120 women will be randomized, in order of recruitment, one by one as control or EVOO groups. EVOO supplementation: The women randomized to EVOO groups will be supplemented daily with 36 mL (three tablespoons) of EVOO with a concentration of phenolic compounds > 500 mg/kg (this concentration of phenols is non-toxic and highly effective, according to the previous reports). The supplementation will start at week 28th of gestation until the term (≥37-weeks), following the published data of our collaborator Dra. Jawerbaum. EVOO will be indicated to be consumed uncooked and within the main meals as reported. All the needed EVOO for the 12 weeks of protocol will be provided monthly to the participants (to assure the correct quality of EVOO).

EXTRA VIRGIN OLIVE OIL CHARACTERIZATION: The EVOO for this project will be obtained from ALONSO (TM), EVOO producers that regularly determine the composition of EVOO, to assure its quality. According to previous publications, the investigators will use EVOO from the varietal Coratina (700 mg/Kg1of polyphenols) that present the higher concentration of phenolic compound compared with other varietals presents in Chile. Considering that the polyphenolic composition of the varietals changes yearly according to the climatological conditions, in collaboration with ALONSO producers, the investigators will measure the lipidic and polyphenol composition, in all the lots of EVOO required for the study.

ADHERENCE AND FOLLOWING: The dietary habits, physical activity, body mass determination and different anthropometric measurements will be obtained by physical examination and questionaries performed at the moment of recruitment and monthly by a nutritionist that support this project and works with Dr. Illanes team in CUA (Dra. Peñailillo). Adherence: Adherence to the supplementation will be evaluated by questionaries. Questionaries: the EVOO consumption will be obtained after application of two nutritional questionaries to determine dietary habits: (1) food frequency questionnaire (FFQ) and (2) mediterranean diet adherence screener (MEDAS), questionary developed and validated for Chilean population by the group of our Co-investigator Dr. Rigotti. The adherence will be considered Good, if questionaries indicated a daily EVOO consumption over 26 g/day, 5 to 7 times per week. As Regular, if daily EVOO consumption was over 26 g/day, but only 3 or 4 times per week, and Bad, if daily EVOO consumption was lower than 26 g/day or lower than 3 times per week. Only Good adherence will be considered for the study. In the sample size determination section, the investigators considered that 25% of recruited women will be lost by low adherences (classified ad regular or bad) as reported in studies of EVOO supplementation.

PARAMETERS TO BE EVALUATED: At the end of pregnancy maternal and umbilical cord blood samples (MPH, MPH + EVOO, MSPH and MSPH + EVOO) will be obtained to evaluate the lipoprotein profile, lipoprotein function, oxidative status, as well as markers of vascular dysfunction.

EXPECTED RESULTS. The aim of this protocol is to determine that the adherence (Good) to the EVOO supplementation protocol will reduce the oxidative status, the markers of inflammation and endothelial dysfunction in the maternal and neonatal blood as well as in placental vessels, promoting an anti-atherogenic lipoprotein profile and function, without reduction of the total cholesterol levels. As a second outcome of this aim, the adherence determination by the dietary questionaries, will also allow to determine the predisposition of this population (pregnant women) to a dietary intervention. This data will be useful to propose bigger interventions in the future. Finally, it is expect to determine the association between EVOO supplementation and clinical parameters of pregnancy outcome (weight gain, blood pressure, birth weight, week of delivery).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 26-28 weeks of gestation
* Singleton pregnancies
* Pregnancies without fetal malformations

Exclusion Criteria:

* Pregnant women with pre-gestational and/or gestational diabetes mellitus
* Pregnant women with obesity before or during pregnancy
* Pregnant women with pre-eclampsia,
* Pregnant women with pregnancy hypertensive syndrome
* Pregnant women with fetal growth retardation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Lipoprotein function | 48 weeks after the end of pregnancy or 60 weeks after randomization
  At the end of pregnancy lipoprotein function determined as conjugated dienes formation (concentration vs time) will be evaluated by ultraviolet absorbance in lipoproteins isolated from maternal and umbilical cord blood
Oxidative status | 48 weeks after the end of pregnancy or 60 weeks after randomization
  At the end of pregnancy oxidative status determined as concentration of oxidized LDL (mg/dL) will be evaluated by ELISA in maternal and umbilical cord blood
Lipid profile | 10 weeks after the end of each pregnancy or 22 weeks after randomization.
  At the end of pregnancy, lipoprotein profile determined as concentration of total cholesterol, LDL, HDL and triglycerides (mg/dL) will be evaluated in the clinical laboratory in maternal and umbilical cord blood

SECONDARY OUTCOMES:
Markers of endothelial dysfunction | 48 week after pregnancy or 60 weeks after randomization
  At the end of pregnancy, markers of endothelial dysfunction determined as levels of soluble VCAM (ng/mL) will be assayed by ELISA in maternal and umbilical blood as well as in placental vessels
Determination of adherence to a mediterranean diet | The adherence to mediterranean diet will be evaluated 4, 8 and 12 weeks after randomization
  Adherence to mediterranean diet, which includes EVOO consumption, will be assayed by the mediterranean diet adherence screener (MEDAS). The adherence will be considered Good, Regular, or Bad according to established and published criteria of MEDAS.
Determination of adherence to EVOO supplementation by food frequency questionnaire | The FFQ will be evaluated 4, 8 and 12 weeks after randomization.
  Adherence to the EVOO supplementation will be evaluated by food frequency questionnaire (FFQ). The adherence will be considered Good, if questionaries indicated a daily EVOO consumption over 26 g/day, 5 to 7 times per week. As Regular, if daily EVOO consumption was over 26 g/day, but only 3 or 4 times per week, and Bad, if daily EVOO consumption was lower than 26 g/day or lower than 3 times per week.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Leiva, PhD, Principal Investigator — Universidad San Sebastian
Locations (1):
- Clinica Universidad de los Andes, Santiago, Las Condes, Chile

IPD SHARING:
Plan to Share IPD: No
The participant will be codified and only clinical parameters are requerid

REFERENCES:
- [Background] Napoli C, Glass CK, Witztum JL, Deutsch R, D'Armiento FP, Palinski W. Influence of maternal hypercholesterolaemia during pregnancy on progression of early atherosclerotic lesions in childhood: Fate of Early Lesions in Children (FELIC) study. Lancet. 1999 Oct 9;354(9186):1234-41. doi: 10.1016/S0140-6736(99)02131-5. PMID 10520631
- [Background] Liguori A, D'Armiento FP, Palagiano A, Balestrieri ML, Williams-Ignarro S, de Nigris F, Lerman LO, D'Amora M, Rienzo M, Fiorito C, Ignarro LJ, Palinski W, Napoli C. Effect of gestational hypercholesterolaemia on omental vasoreactivity, placental enzyme activity and transplacental passage of normal and oxidised fatty acids. BJOG. 2007 Dec;114(12):1547-56. doi: 10.1111/j.1471-0528.2007.01510.x. Epub 2007 Sep 27. PMID 17903226
- [Background] Leiva A, de Medina CD, Salsoso R, Saez T, San Martin S, Abarzua F, Farias M, Guzman-Gutierrez E, Pardo F, Sobrevia L. Maternal hypercholesterolemia in pregnancy associates with umbilical vein endothelial dysfunction: role of endothelial nitric oxide synthase and arginase II. Arterioscler Thromb Vasc Biol. 2013 Oct;33(10):2444-53. doi: 10.1161/ATVBAHA.113.301987. Epub 2013 Aug 15. PMID 23950140
- [Background] Guasch-Ferre M, Li Y, Willett WC, Sun Q, Sampson L, Salas-Salvado J, Martinez-Gonzalez MA, Stampfer MJ, Hu FB. Consumption of Olive Oil and Risk of Total and Cause-Specific Mortality Among U.S. Adults. J Am Coll Cardiol. 2022 Jan 18;79(2):101-112. doi: 10.1016/j.jacc.2021.10.041. PMID 35027106
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Gomez Ribot D, Diaz E, Fazio MV, Gomez HL, Fornes D, Macchi SB, Gresta CA, Capobianco E, Jawerbaum A. An extra virgin olive oil-enriched diet improves maternal, placental, and cord blood parameters in GDM pregnancies. Diabetes Metab Res Rev. 2020 Nov;36(8):e3349. doi: 10.1002/dmrr.3349. Epub 2020 Jun 24. PMID 32447799